CLINICAL TRIAL: NCT03062371
Title: Measuring the Feasibility and Preliminary Efficacy of Therapeutic Playgroups in Early Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Florida Gulf Coast University (Other)
Responsible Party: Principal Investigator, Dr. Sarah Fabrizi, Principal Investigator, Florida Gulf Coast University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-22
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Developmental Delay
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Playgroup Intervention (Experimental): The approach of the playgroup is to promote healthy family play routines with an emphasis on child and family well-being. The intervention types for playgroup sessions included the occupation of play, activities to promote play and participation, educating caregivers through modeling and coaching, advocating for the child and family, and the use of group sessions. Specific playgroup strategies included a predictable routine, following the child's lead, imitating the child, modeling of new behaviors, and scaffolding play - within both the social and physical environment. When developing activities, play objects that families have at home and are easily obtained were used and positioned intentionally with respect to the child-caregiver dyad and the group as a whole.
  Interventions: Behavioral: Playgroup

INTERVENTIONS:
Behavioral: Playgroup — A semi-structured gathering of caregivers and their children in a community setting developed and implemented by a skilled provider.
  Other Names: community playgroup, developmental playgroup

SUMMARY:
Play builds social-emotional skills. Therapeutic playgroups facilitate parent-child interaction these and provide opportunities for parents to engage with their children and other adults and learn more about development.

Objective: The purpose of this research is to investigate if children between the ages of 15 months and 5 years old, with and without special needs, demonstrate improved levels of playfulness and social- emotional growth after participation in a therapeutic playgroup, provided in various settings in the community. Investigators will also examine the impact that these playgroups have on participating caregiver's confidence and competence.

Method: A quasi-experimental mixed methods sequential explanatory design will be used. The Test of Playfulness will measure child playfulness, the Social Profile and Assessment of Preschool Children's Participation play sub scale will determine child participation, the Devereux Early Childhood Assessment will determine social emotional growth, and the Parenting Sense of Competence Scale will determine the caregiver sense of competence. Mean differences will be analyzed using a mixed analysis of variance to determine significant changes over time for each group. Follow up surveys with parents and providers will determine parent perception of playgroup and provider perception of effectiveness and feasibility. We hypothesize that playgroups will have a significant effect on child playfulness, social-emotional growth, participation, and parent competence. We also hypothesize that participating parents will report benefits of playgroups and providers will share benefits and barriers to including therapeutic playgroups as part of comprehensive early intervention services.

DETAILED DESCRIPTION:
All children have the right to play; the right to play is enshrined in Article 31 of the UN Convention on the Rights of the Child. Play is the fundamental way that children enjoy their childhood. It is essential to their quality of life as children.

Play permits children to engage and interact with the world around them. This exploration supports the development of their social and cognitive skills needed for learning. Research has described play as the most important 'work' a child engages him or herself in. Children with developmental disabilities often have difficulties establishing peer relations. Impairments in social competence can have adverse effects on play and can result in negative behaviors that are detrimental to forming relationships. As a result, the purpose of this research study is to determine if an intervention playgroup will increase playfulness and social participation for children ages 18 months to five years. The current research will also measure parental confidence in its attempt to understand the full effect of playgroups on the family unit.

Playgroups have the potential to encourage parents, caregivers, and their children to play and have fun together safely. Playgroups offer a stimulating environment that facilitates a child's developmental needs and encourages parents to develop stable support networks. According to research, to enhance participation for children with disabilities, play must be involved in something or with someone, must offer a sense of inclusion, must have choice or control in the activity, and must be working towards a goal or enhancing the child's quality of life.

Early intervention involves establishing developmentally appropriate play as an outcome or means to achieve goals. Playgroups have the added benefit of allowing the opportunity to coach caregivers on parenting, creating social networks, forging friendships, and seeking community connectedness. Practitioners who use a family centered approach see significant improvements in both occupational performance and parent confidence . Carryover of skills from the playgroup and into the home will be accomplished through the interaction between dyads. Findings from the National Early Intervention Longitudinal Study (NEILS) showed that 98% of families participating in early intervention felt competent in caring for their children's basic needs and 90% reported that early intervention services had improved their ability to help their children develop and learn.

Playfulness is defined as the way in which the child approaches any activity or task. Arguably, playfulness can be considered more important to defining play than the play activity itself. There is a strong correlation between playfulness and coping strategies a child will use later in life. Play positively affects cognition and problem-solving, thereby increasing their coping abilities. Through play, a child develops strategies of managing and exploring a world of rich interactions.

Currently, there are limited studies describing the effectiveness of playgroups on a child's playfulness and social participation. Countries such as England and Australia have both local and national playgroup associations with established procedures for organizing and running a group headed by a team of professional coordinators. However, in the US, playgroups are sparse, less formal, and receive little to no support from national or state associations. There is a need for future research to explore the benefits of playgroups within the local community to remedy the lack of support in the US and provide an adequate play environment to children of any developmental background.

Major Research questions:

Will children ages 15 months to five years demonstrate increased playfulness and social participation after participating in playgroup? Will the caregiver of a child ages 18 months to five years report increased confidence in community outings with their child? Will providers identify benefits and barriers to providing therapeutic playgroups as part of early intervention services?

Hypothesis:

Children that participate in playgroups will show increased playfulness and social participation. Their primary caregiver will report increased confidence in community outings with their child.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers and children ages 15 months to 5 years old
* At least one caregivers must be able to attend all playgroup sessions

Exclusion Criteria:

-Caregivers must speak English or provide translator

Ages: 15 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Social Emotional status using the Devereux Early Childhood Assessment, a parent report | change - week 1 and week 8
  Use of t-score

SECONDARY OUTCOMES:
Parent Competence/ Efficacy , a Likert scale parent report | change - week 1 and week 8
  Parent report of efficacy in their role, efficacy scale is reverse coded to combine to form a total score for parent competence, higher score indicates higher level of competence
Participation | change - week 1 and week 8
  Young Child Participation and Environment Measure (YC-PEM)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Fabrizi, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Sarah Fabrizi, Fort Myers, Florida, United States

REFERENCES:
- [Background] Andrews F, Griffiths N, Harrison L, Stagnitti K. Expectations of parents on low incomes and therapists who work with parents on low incomes of the first therapy session. Aust Occup Ther J. 2013 Dec;60(6):436-44. doi: 10.1111/1440-1630.12044. Epub 2013 Jun 18. PMID 24299483
- [Background] Bundy, A. (2010). Test of playfulness (ToP) 4.2 manual revised 11/10. Lidcombe, Australia: University of Sydney.
- [Background] Cameron D, Leslie M, Teplicky R, Pollock N, Stewart D, Toal C, Gaik S. The clinical utility of the test of playfulness. Can J Occup Ther. 2001 Apr;68(2):104-11. doi: 10.1177/000841740106800206. PMID 11355615
- [Background] Case-Smith J. Systematic reviews of the effectiveness of interventions used in occupational therapy early childhood services. Am J Occup Ther. 2013 Jul-Aug;67(4):379-82. doi: 10.5014/ajot.2013.007872. No abstract available. PMID 23791311
- [Background] Donohue, M.V. (2013). Social profile: Assessment of social participation in children, dolescents, and adults. Retrieved from http://myaota.aota.org/shop_aota/prodview.aspx?TYPE=D&PID=160964175&SKU=124 4
- [Background] Ginsburg KR; American Academy of Pediatrics Committee on Communications; American Academy of Pediatrics Committee on Psychosocial Aspects of Child and Family Health. The importance of play in promoting healthy child development and maintaining strong parent-child bonds. Pediatrics. 2007 Jan;119(1):182-91. doi: 10.1542/peds.2006-2697. PMID 17200287
- [Background] Graham F, Rodger S, Ziviani J. Effectiveness of occupational performance coaching in improving children's and mothers' performance and mothers' self-competence. Am J Occup Ther. 2013 Jan-Feb;67(1):10-8. doi: 10.5014/ajot.2013.004648. PMID 23245778
- [Background] Hoogsteen L, Woodgate RL. Can I play? A concept analysis of participation in children with disabilities. Phys Occup Ther Pediatr. 2010 Nov;30(4):325-39. doi: 10.3109/01942638.2010.481661. PMID 20735196
- [Background] Johnston, C., & Mash, E.J. (1989). A measures of parenting satisfaction and efficacy. Journal of Clinical Child Psychology, 18,167-175. Retrieved from https://researchingparents.wordpress.com/2013/02/15/parenting-sense-of-competence- psoc/
- [Background] Mize, J., & Pettit G.S. (2010). The mother-child playgroup as socialisation context: a short-term longitudinal study of mother-child-peer relationship dynamics. Early Child Development and Care, 180(10), 1271-1284. DOI: 10.1080/0300443090298147
- [Background] O'Brien J, Coker P, Lynn R, Suppinger R, Pearigen T, Rabon S, St Aubin M, Ward AT. The Impact of Occupational Therapy on a Child's Playfulness. Occup Ther Health Care. 2000;12(2-3):39-51. doi: 10.1080/J003v12n02_03. PMID 23951988
- [Background] Strange C, Fisher C, Howat P, Wood L. Fostering supportive community connections through mothers' groups and playgroups. J Adv Nurs. 2014 Dec;70(12):2835-46. doi: 10.1111/jan.12435. Epub 2014 May 7. PMID 24805198
- [Background] Saunders I, Sayer M, Goodale A. The relationship between playfulness and coping in preschool children: a pilot study. Am J Occup Ther. 1999 Mar-Apr;53(2):221-6. doi: 10.5014/ajot.53.2.221. PMID 10200846
- [Background] Vedeler, L. (2004). Social coping strategies in pre-school play. How do children with disabilities succeed in play groups with other children? Scandinavian Journal of Disability Research, 6(3), 192-205, DOI: 10.1080/15017410409512652